CLINICAL TRIAL: NCT02696070
Title: A Multi-Center, Randomized, Sham-Controlled, Double-Blind Study of Pulsed Electromagnetic Field (PEMF) Therapy to Evaluate Small Fiber Nerve Growth and Function in Subjects With Painful Peripheral Diabetic Neuropathy
Brief Title: Nociceptive Pain Fiber Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenesis Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBI.2015.002
Record Dates: First submitted 2016-02-17; First posted 2016-03-02 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2016-12

CONDITIONS: Painful Peripheral Diabetic Neuropathy
Keywords: Pain; Diabetic Neuropathy; Pulsed Electromagnetic Energy Field; PEMF; PPDN
MeSH Terms: conditions — Pain; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham of Provant (Other): Sham of Provant
  Interventions: Device: Provant Therapy System
- Active Treatment (Other): Active Provant Treatment
  Interventions: Device: Provant Therapy System

INTERVENTIONS:
Device: Provant Therapy System

SUMMARY:
This study is designed to evaluate the effectiveness of the Provant Therapy System in improving localized nerve growth and skin perfusion in subjects with painful peripheral diabetic neuropathy of the foot.

DETAILED DESCRIPTION:
The study is multi-site, randomized, double-blind, sham-controlled study of the safety and efficacy of multi-dose Provant therapy to evaluate neuronal and vascular response in the treatment of subjects with painful peripheral diabetic neuropathy. Subjects will be randomized in a 2:1 ratio to receive therapy with an active device or an identical inactive sham device. Subjects will treat at home twice daily for 60 days after which they will return to the clinic for final evaluations. Subjects will be evaluated at the research center for a Baseline/Enrollment visit and again at Day 61 where assessments for safety, concomitant medications, Sympathetic Skin Response (SSR), Nerve Conduction Velocity (NCV), Skin Perfusion Pressures (SPP), and Skin Biopsy will be completed. Subjects will be contacted via telephone at Day 14, Day 28 and Day 42 to assess adherence, safety, and concomitant medications. Subjects will also complete a Response to Study Device form which will capture their daily pain score.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age is greater than or equal to 22 years and less than 80 years of age.
2. Subject has documented Type 2 diabetes.
3. Subject has an HgbA1c > 7% and < 10%.
4. Subject has peripheral diabetic neuropathy with pain, numbness, tingling, and/or burning in at least one foot confirmed by a positive provocative sign and a positive Tinel's sign. If both feet are involved, the one with the greatest severity will be selected as the index foot.
5. Subject is in pain Phase 2, 3, or 4 (Appendix C).
6. Subject is willing and able to give written informed consent and to comply with all parts of the study protocol including diary entries.
7. Female subjects must be post-menopausal, surgically sterile, abstinent, or practicing (or agree to practice) an effective method of birth control if they are sexually active for the duration of the study. (Effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier methods, and/or male partner sterilization).

Exclusion Criteria:

1. Subject has Type 1 diabetes.
2. Subject is in pain Phase 1 or 5 (Appendix C).
3. Subject has an active, open ulcer on either lower extremity of arterial, venous or mixed disease origin.
4. Subject has peripheral arterial disease as determined by an Ankle-Brachial Index (ABI) of >1.40 or < 0.80. See Appendix E for details on obtaining the ABI.

   NOTE: If the difference in the brachial pulse pressure between the right and left arms is > 10 mmHg, the subject will not be eligible for enrollment and will be referred to a cardiologist for further evaluation.
5. Subject has venous insufficiency classified by the Venous Insufficiency Classification System (CEAP) of grades C3, C4, C5, or C6. See Appendix F for description of the venous insufficiency grading.
6. Subject has undergone decompression surgery on the index foot to treat peripheral neuropathy within 2 years of the Screening Visit.
7. Subject requires or anticipates the need for surgery of any type during the 60 day treatment period.
8. Subject is a smoker or has been a smoker within one year of the Screening Visit.
9. Subject has a total foot thickness (plantar surface to mid-dorsal surface) of > 6 centimeters.
10. Subject anticipates travelling over the course of the 60 day treatment period.
11. Subject has received any investigational drug or device within 30 days or 5 half-lives of the drug, whichever is longer, prior to the Screening Visit or is enrolled in another clinical trial.
12. Subject has undergone any local injection into the index foot within 30 days prior to the Screening Visit or within 6 weeks prior to the Screening Visit for long acting lidocaine injection products.
13. Subject has used systemic corticosteroids within 2 months of the Screening Visit.
14. Subject has a history of any uncontrolled medical illness that in the investigator's judgment places the subject at unacceptable risk for receipt of PEMF therapy.
15. Subject has a history of malignancy within the past five years other than successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin in the treatment area and/or localized in situ carcinoma of the cervix.
16. Subject has a serious psychosocial co-morbidity.
17. Subject has a history of drug or alcohol abuse, as confirmed by urine drug screen, within one year prior to the Screening Visit.
18. Subject has an implanted pacemaker, defibrillator, neurostimulator, spinal cord stimulator, bone stimulator, cochlear implant, or other implanted device with an implanted metal lead(s).
19. Subject is currently pregnant or planning on becoming pregnant prior to Day 60.
20. Subject has been previously treated with the PROVANT Therapy System.
21. Subject is unwilling or unable to follow study instructions, or comply with the treatment regimen and study visits.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Extremity Health Center, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham of Provant: Inactive / sham Provant Therapy System. Subjects were instructed to treatment with an inactive Provant Therapy Unit that did not emit a pulsed electromagnet field.
- Active Treatment: Acitve Provant Therapy System. Subjects were instructed to treatment with an active Provant Therapy Unit that emitted a pulsed electromagnet field.
Period: Overall Study
Arm/Group | Sham of Provant | Active Treatment
Started | 8 | 14
Completed | 7 | 12
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham of Provant | Active Treatment | Total
Number analyzed (Participants) | 8 | 14 | 22
Age, Continuous [Mean (Full Range); unit: Years] | 62.14 [56 to 76] | 59 [46 to 74] | 60.14 [46 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 12 | 19
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: Count of Participants]
  United States | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Changes in Small Nerve Fiber Density by Assessment of a Skin Biopsy Comparing Baseline to Day 60
Description: The mean percent change in intraepidermal nerve fiber density mean values for mean nerve fibers per millimeter squared from baseline to Day 60 was calculated for each treatment group (value at 60 days minus value at baseline).
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: nerve fibers / mm squared
Arm/Group | Sham of Provant | Active Treatment
Number analyzed (Participants) | 7 | 12
nerve fibers / mm squared | .1 (.53) | .1 (.45)

ADVERSE EVENTS:
Arm/Group | Sham of Provant | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/14
Other Adverse Events (participants affected / at risk) | 0/8 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication Rights. Independent analysis and/or publication of data generated or arising from the performance of this Agreement is not permitted without the prior written consent of Regenesis. Such consent may be contingent on Regenesis' review and approval of any proposed analysis and manuscript. Institution will retain the right to review and analyze the database created from this study for its own scientific purposes so long as such scientific purposes are non-commercial in nature.